CLINICAL TRIAL: NCT05274243
Title: 2-HOBA Phase 2 Clinical Trial in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michelle Ormseth, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 220141
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 2-(aminomethyl)phenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2-HOBA (Experimental): 2-HOBA acetate (2-Hydroxybenzlamine acetate) 750mg (provided as three 250mg capsules) three times per day for 4 weeks
  Interventions: Drug: 2-HOBA
- Placebo (Placebo Comparator): Matching placebo (provided as three capsules) three times per day for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2-HOBA — 2-HOBA acetate (2-Hydroxybenzlamine acetate) 750mg (provided as three 250mg capsules) three times per day for 4 weeks
  Other Names: 2-hydroxybenzylamine; salicylamine; IUPAC name: 2-(aminomethyl)phenol
  Arms: 2-HOBA
Other: Placebo — Placebo (provided as three capsules) three times a day for 4 weeks
  Arms: Placebo

SUMMARY:
This is a phase 2 study to determine 2-HOBA's tolerability, safety, and effect on isoLG-adducts in patients with rheumatoid arthritis (RA) patients. Up to 32 subjects will be randomized to 750mg 2-HOBA or matching placebo three times a day for 4 weeks.

As primary outcome measures investigators will compare tolerability and adverse events and changes in isoLG adducts in active and placebo arms. Among prespecified exploratory outcomes investigators will compare changes in markers of inflammation, DAS28 score, and 24-hour blood pressure in active and placebo arms. This pilot study will inform the feasibility and design of future studies to examine the efficacy of 2-HOBA in RA patients.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic inflammatory autoimmune disease affecting 1% of the population. Aggressive treatment is a fundamental therapeutic strategy to improve disease-related outcomes and cardiovascular disease, which contributes to excess mortality in RA. Thus, therapeutics targeting novel pathways that treat RA and reduce cardiovascular risk are needed. A potential target is blocking the proinflammatory, immunogenic, and proatherogenic consequences of isolevuglandins (isoLGs).

IsoLGs are highly reactive dicarbonyl products of oxidative stress that bind covalently to proteins causing conformational changes rendering them immunogenic and proinflammatory. Two decades of work at Vanderbilt led to the identification of 2-hydroxybenzylamine (2-HOBA) as a highly effective scavenger of reactive dicarbonyls such as isoLGs. Scavenging reactive dicarbonyls is preferable to using antioxidants because reactive oxygen species are necessary for normal cellular function. In animal models of autoimmunity, hypertension, and atherosclerosis 2-HOBA reduced inflammation, autoantibodies, blood pressure, and atherosclerosis, and in human phase 1 clinical studies in healthy volunteers 2-HOBA was well tolerated.

In this phase 2 study investigators will randomize up to 32 subjects with RA meeting inclusion/exclusion criteria to 750mg 2-HOBA or matching placebo three times a day for 4 weeks. Randomized subjects will have study visits at week 0 and week 4. At each visit a history and physical exam with joint counts, questionnaire, blood draw and 24-hour blood pressure will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Meets 2010 American College of Rheumatology/European League Against Rheumatism Rheumatoid Arthritis classification criteria
* ≥ 4 tender or swollen joints
* No change in DMARDs, glucocorticoids in ≥ 4 weeks
* If of childbearing potential, willingness to use effective birth throughout study and 4 weeks after completion of the study (examples: condom, diaphragm, oral contraceptive pill, intrauterine device)
* If using non-steroidal anti-inflammatory drugs (NSAIDs), willingness to discontinue use of NSAIDs for 2 weeks prior to the study and throughout the study

Exclusion Criteria:

* Pregnant or breastfeeding
* Active cancer except non-melanoma skin cancer
* Active infection
* Concomitant inflammatory autoimmune disease
* Major surgery in ≤ 3 months
* Aspirin allergy
* Use of MAO-I
* Estimated creatinine clearance <30 ml/min
* Prior diagnosis of liver cirrhosis or the following abnormal liver function studies: AST or ALT >1.5x the upper limit of normal or total bilirubin ≥1.5 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability (adverse events) | Baseline to 4 weeks
  Rates of adverse events will be compared between active and placebo arms and presented as summary statistics.
Cellular isolevuglandin (isoLG) adducts | Baseline to 4 weeks
  Change in percentage of cellular isoLG adducts will be compared between active and placebo arms.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ormseth, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified data will be available upon reasonable written request in conjunction with appropriate data use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication and for 1 year.
Access Criteria: Only deidentified data will be available upon reasonable written request in conjunction with appropriate data use agreement. Interested parties may contact the study PI.

DOCUMENTS (1):
  • Informed Consent Form (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/43/NCT05274243/ICF_000.pdf